CLINICAL TRIAL: NCT06113224
Title: Characterization of Anti-HLA Alloimmunization After Pulmonary Valve Homograft Insertion (CAssIOPé)
Brief Title: Characterization of Anti-HLA Alloimmunization After Pulmonary Valve Homograft Insertion
Acronym: CAssIOPé
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM22_0448
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Lung Graft Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control patients (Active Comparator): Patients with an indication for cardiac surgery with extracorporeal circulation but without homograft
  Interventions: Procedure: Blood collection T0; Procedure: Blood collection 6 months
- Lung homograft patients (Experimental): patients requiring lung homograft implantation
  Interventions: Procedure: Blood collection T0; Procedure: Blood collection 6 months

INTERVENTIONS:
Procedure: Blood collection T0 — 2 blood samples will be taken in addition to the pre-operative check-up.
Procedure: Blood collection 6 months — 1 blood sample will be taken 6 months after surgery.

SUMMARY:
This is a prospective, monocentric, observational cohort study whose main objective is to describe the number and rate of patients who developed DSAs (Donor Specific Antibody) at 6 months post-surgery with implantation of a cryopreserved lung homograft.

DETAILED DESCRIPTION:
Lung homograft is used in a large number of complex malformations. It is accepted that homografts may induce immune reactions in the recipient, but no immunological studies have been carried out to characterize the recipient's immune reactions to the homograft and their potential impact on valve function. In this project, the authors propose to study the immunizing character of cryopreserved lung homografts by identifying the appearance of antibodies directed against the HLA, DSA (Donor Specific Antibodies) molecules of the graft (lung homograft) at 1 month and 6 months after its surgical implantation.The primary objective will be analyzed by describing the rate of patients who developed DSA at 6 months post-surgery with implantation of a cryopreserved lung homograft.

ELIGIBILITY:
Inclusion Criteriafor control patients:

* Patient receiving a cryopreserved pulmonary valve homograft
* Patient aged 14 or over
* Signature of consent by adult patients/parents/guardians and assent by children

Inclusion Criteriafor patients with lung homograft :

* Patientsreceiving a cardiac surgery with extracorporeal circulation and without lung homograft

Exclusion Criteria for both group

* Emergency surgery patient
* Pregnant women or childbirth within the last 6 months
* Transfusion during the surgery or within the last 6 months
* Patient with DSAs detected before the surgery
* Patient with anti-HLA antibodies (non-DSAs) detected before the surgery

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Detection of DSA at 6 months | 6 months
  Luminex® detection of DSA at 6 months after lung homograft implantation

SECONDARY OUTCOMES:
DSA Quantification | 6 months
  DSA will be quantified in patients who developed DSA 6 months after lung homograft implantation
antibody anti-HDLA (non DSA) detection | 6 months
  Detection or non-detection of non-DSA anti-HLA antibodies will be assessed by Mean Fluorescence Intensity.
Early degeneration of the homograft | 6 months
  The early degeneration of the homograft will be defined by the occurrence of at least one of the following criteria:
  * Need to replace lung homograft
  * Need for dilatation during catheterization of lung homografts
  * Maximum gradient across the lung homograft ≥ 30mmhg on echography at 6 months
  * Pulmonary insufficiency ≥ moderate on echography at 6 months